CLINICAL TRIAL: NCT04177615
Title: Randomized Assessment of Rapid Endovascular Treatment in Basilar Artery Occlusion Stroke in 115 Hospital
Acronym: RARETBAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Tran Nguyen Uyen Dung, Randomized Assessment of Rapid Endovascular Treatment in Basilar Artery occlusion stroke in 115 hospital, University of Medicine and Pharmacy at Ho Chi Minh City
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: yds2019
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Stroke, Acute; Basilar Artery Occlusion
Keywords: Ischemic stroke; Basilar Artery Occlusion
MeSH Terms: conditions — Stroke; Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thromboectomy and rTPA (Experimental): use thromboectomy and rtpa for patient with basilar artery occlusion stroke in 24 hour
  Interventions: Procedure: Thromboectomy
- rTPA( recombinant tissue plasminogen activator ) (No Intervention): use rtpa for patient with basilar artery occlusion stroke in 24 hour

INTERVENTIONS:
Procedure: Thromboectomy — Thromboectomy in Basilar Artery Occlusion patients
  Arms: Thromboectomy and rTPA

SUMMARY:
This is a prospective, open lable studies conducted in 115 hospital to compare between thromboectomy and Recombinant Tisue Plasminogen Activator only to evaluate the eficacy and safety of endovascular treatment in basilar artery occlusion stroke patients

DETAILED DESCRIPTION:
Acute basilar artery thrombosis is associated with a poor prognosis. Prevalence of basilar artery occlusion are not known. Although basilar artery occlusion has been reported in 2 per 1000 autopsy cases, basilar artery thrombosis may, in stroke registries, explain as many as 27% of ischemic strokes occurring in the posterior circulation.Various treatments were tried in groups of patients with vertebrobasilar territory infarction but evidence based was not cleared previous studies. Therefore, we conduct this study to evaluate the eficacy and safety of endovascular treatment in basilar artery occlusion stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Patients admit to 115 hospital in 24h of Basilar Artery Occlusion Stroke
* NIHSS > 4 points

Exclusion Criteria:

* Patients refuse to participate in studies
* Patients with contraindication of either rTPA or thromboectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2019-11-19 (Estimated); Primary Completion 2020-11-19 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
NIHSS in patients wtih Basilar Artery Occlusion Stroke after 24hour admission | 24 hours from admission
  NIHSS in patients wtih Basilar Artery Occlusion Stroke after 24hour admission
Survival rate in patients with Basilar Artery Occlusion Stroke | 3 months from admission
  Survival rate in patients with Basilar Artery Occlusion Stroke

SECONDARY OUTCOMES:
mRS in patients with Basilar Artery Occlusion Stroke | 3 months from admission
  mRS in patients with Basilar Artery Occlusion Stroke

CONTACTS AND LOCATIONS:
Overall Officials: TUAN D Tran, MD, Study Chair — UMP university

IPD SHARING:
Plan to Share IPD: No